CLINICAL TRIAL: NCT02927171
Title: Shifting Rehabilitation Paradigms in Skilled Nursing Facilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: E2193-P; I21RX002193 (NIH)
Record Dates: First submitted 2016-09-26; First posted 2016-10-06 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Physical Deconditioning
Keywords: Skilled Nursing Facility; Post-Acute Care; Older Adults; Physical Function; Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Skilled nursing facility rehabilitation therapists provide all patients with usual standard of care.
- I-STRONGER (Experimental): IntenSive Therapeutic Rehabilitation for Older Skilled NursinG HomE Residents (I-STRONGER) Progressive, high-intensity strengthening and functional interventions to facilitate independence with functional activities. Skilled nursing facility rehabilitation therapists will be trained in I-STRONGER intervention and will implement to all eligible patients as new standard of care.
  Interventions: Other: IntenSive Therapeutic Rehabilitation for Older Skilled Nursing Home Residents

INTERVENTIONS:
Other: IntenSive Therapeutic Rehabilitation for Older Skilled Nursing Home Residents — Progressive, high-intensity strengthening and functional interventions to facilitate independence with functional activities.
  Other Names: I-STRONGER
  Arms: I-STRONGER

SUMMARY:
This study seeks to improve rehabilitation methods for restoring physical function with skilled nursing facility care. More specifically, this study is designed to evaluate the effectiveness of an intensive therapeutic rehabilitation program for older adult skilled nursing home residents compared to usual care.

DETAILED DESCRIPTION:
There is growing recognition that acute hospitalization contributes to marked functional decline in older adults. Nearly 20% of all hospitalized older adults are discharged to a skilled nursing facility (SNF) to address these functional deficits. However, rehabilitation in SNFs may not adequately restore physical function, which potentially contributes to poor community discharge rates. Strikingly, only 37% of all patients admitted to SNFs are discharged to a community setting, which suggests a paradigm shift is required to optimize rehabilitation within SNFs. Currently, usual care rehabilitation in SNFs consists of low-intensity rehabilitation interventions, which are physiologically inadequate to induce meaningful changes in skeletal muscle strength and physical function. Therefore, the investigators propose a novel "IntenSive Therapeutic Rehabilitation for Older skilled NursinG HomE Residents" (I-STRONGER) program, which integrates principles of physiologic tissue overload into combined strengthening and functional interventions for greater gains in physical function. The overall goals of this investigation are to 1) demonstrate feasibility of I-STRONGER in SNF settings and 2) determine the effectiveness of I-STRONGER in improving physical function. A comparison of usual care (UC) with I-STRONGER will occur using a staged, 2 group design (independent cohorts), with a single SNF serving as its own control. The first cohort of SNF patients will participate in UC (Stage 1) and after therapist training on ISTRONGER is completed, a second cohort of patients entering the same facility will participate in I-STRONGER (Stage 2). The feasibility of I-STRONGER will be evaluated by patient acceptability and therapist compliance measures. Sample size estimates (using patients with mobility deficits in home health settings) suggest at least 86 participants are necessary to be adequately powered. Heterogeneity of the sample will be re-evaluated during the study period using SNF data and sample size estimates may be adjusted as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 years of age who are admitted to a skilled nursing facility following hospitalization
2. Qualify to receive at least physical therapy services

Exclusion Criteria:

* Patients with primary diagnoses related to neurological disorders will be excluded as patient needs require more of a motor control approach rather than the proposed high-intensity approach. Such patient populations include:

  * Parkinson's Disease
  * Traumatic Brain Injury
  * Recent Cerebral Vascular Accident
  * Alzheimer's Disease
* Patients on hospice care will be excluded as the approach is based on palliative principles.
* Other patients to be excluded will include those with conditions where strength training is contraindicated (as indicated by the American College of

Sports Medicine Guidelines for Exercise Testing and Prescription):

* Recent unstable fracture
* Advanced congestive heart failure
* Bone metastasis sites
* Tumors in strengthening target areas
* Acute Illness
* Recent myocardial infarction (within 3-6 weeks)
* Weight bearing restrictions on graft or fracture sites
* Exposed tendon or muscle
* Absence of pedal pulses
* Presence of fistula
* Platelet levels <50,000/ L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-02-28 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E. Stevens-Lapsley, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (3):
- United States (3):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Community Living Center, Aurora, Colorado
  - Brookdale Senior Living, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mallinson T, Deutsch A, Bateman J, Tseng HY, Manheim L, Almagor O, Heinemann AW. Comparison of discharge functional status after rehabilitation in skilled nursing, home health, and medical rehabilitation settings for patients after hip fracture repair. Arch Phys Med Rehabil. 2014 Feb;95(2):209-17. doi: 10.1016/j.apmr.2013.05.031. Epub 2013 Jul 10. PMID 23850612
- [Result] Peterson MJ, Crowley GM, Sullivan RJ, Morey MC. Physical function in sedentary and exercising older veterans as compared to national norms. J Rehabil Res Dev. 2004 Sep;41(5):653-8. doi: 10.1682/jrrd.2003.09.0141. PMID 15558394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a skilled nursing facility between the dates of 02.28.2016 and 10.30.2018
Pre-assignment Details: There were no exclusions of participants. All eligible, willing participants were allocated to one of two arms.
Period: Overall Study
Arm/Group | Usual Care | I-STRONGER
Started | 53 | 51
Completed | 53 | 50
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: 1 participant in the I-STRONGER arm was lost to follow-up. They were discharged home early, and discharge outcomes were not assessed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | I-STRONGER | Total
Number analyzed (Participants) | 53 | 50 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.0 (9.6) | 77.3 (10.8) | 77.65 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 44 | 48 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 51 | 43 | 94
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 12 | 28
  White | 34 | 31 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 7 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Short Physical Performance Battery (SPPB)
Description: Global measure of lower extremity function, which consists of walking speed, chair stands, and balance tests. Minimum scores are 0 and maximum scores are 12. Higher scores indicate better function.
Time Frame: Change from SNF Admission to SNF Discharge (Expected average length of stay: 21 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | I-STRONGER
Number analyzed (Participants) | 53 | 50
score on a scale | 3.6 (2.3) | 4.3 (2.7)
Statistical Analysis 1: Comparison: Usual Care; Test type: Other; p = 0.17, t-test, 1 sided

2. Secondary Outcome: Gait Speed
Description: Time it takes to walk a 4 meter path. Lower scores indicate better function.
Time Frame: Change from SNF Admission to SNF Discharge (Expected average length of stay: 21 days)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Usual Care | I-STRONGER
Number analyzed (Participants) | 53 | 50
seconds | 0.3 (0.2) | 0.5 (0.3)

3. Other Pre Specified Outcome: Patient Satisfaction Survey
Description: 8 Question survey, scoring each questions on a 1-10 scale (1=not at all, 10=extremely). Higher scores indicate higher satisfaction.
Time Frame: Quantification at SNF Discharge (Expected average length of stay: 21 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | I-STRONGER
Number analyzed (Participants) | 53 | 50
score on a scale | 54.6 (7.9) | 59.4 (7.3)

ADVERSE EVENTS:
Time Frame: Baseline through discharge from Skilled Nursing Facility (average 21 days)
Arm/Group | Usual Care | I-STRONGER
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/50
Other Adverse Events (participants affected / at risk) | 0/53 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT02927171/Prot_SAP_000.pdf